CLINICAL TRIAL: NCT04624022
Title: Evaluation of Implanted Perforated Lacrimal Punctal Plugs Using Anterior Segment Optical Coherence Tomography.
Brief Title: AS OCT Evaluation for Perforated Punctual Plugs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Heba Radi AttaAllah, Assistant prof of Ophthalmology, Minia University
Other Study IDs: 620-5/2020
Record Dates: First submitted 2020-10-29; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Punctal Stenosis
Keywords: Punctual stenosis; Perforated Lacrimal Punctal Plugs; AS-OCT

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Anterior segment optical coherent tomography — Examination of the implanted perforated lacrimal plugs using anterior segment optical coherent tomography

SUMMARY:
Evaluation of the perforated punctal plugs after implantation in cases of punctal stenosis regarding position and patency in the early postoperative period (during the first operative weak)

DETAILED DESCRIPTION:
Prospective non randomized case series study included 50 eyes. The study is conducted on patients attending to the oculoplastic unit of ophthalmology department of Minia university hospital. Informed consents were obtained from the participants in this study. The study was adherent to the tenets of declaration of Heleniski.

Anterior segment optical coherence tomography(AS-OCT) was performed for the included patients after perforated plug implantation (during the first operative weak)

ELIGIBILITY:
Inclusion Criteria:

* Patients with punctal stenosis who will be treated by implantation of perorated punctal plugs

Exclusion Criteria:

* Patients who are not willing to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with epiphora will be evaluated to exclude other causes than punctal stenosis. Perforated punctal plugs were implanted under topical anaesthesia. patients follow up and AS-OCT
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-11-05 (Estimated); Study Completion 2020-11-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the fitting of implanted perforated lacrimal plugs | first week post-operatively
  Either plug is in place or rotated
Evaluation of the patency of the plugs | first week post-operatively
  Either plug is patent or occluded
Evaluation any contents within the plugs | first week post-operatively
  Blood/ Tears/ Debris
Evaluation of the lower tear film height | first week post-operatively
  measuring the tear film meniscus height at the lower lid margin (at the centre of the inferior limbus), height is measured in micrometers
Evaluation of the tear level within the plug | first week post-operatively
  Either within the lower half or upper half of the plug

CONTACTS AND LOCATIONS:
Overall Officials: Heba AttaAllah, MD, Principal Investigator — Faculty of Medicine, Minia University
Locations (1):
- Ophthalmology department/ Minia University Hospital/Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdallah RMA, Elshafei AMK, AttaAllah HR. Evaluation of implanted perforated lacrimal punctal plugs using anterior segment optical coherence tomography. Eye Vis (Lond). 2021 Oct 3;8(1):36. doi: 10.1186/s40662-021-00259-x. PMID 34600582